CLINICAL TRIAL: NCT04793399
Title: Multicenter, Open-label, Phase Ib/II Trial to Evaluate Safety and Efficacy for the Combination of Bosutinib Plus Atezolizumab in Newly Diagnosed Chronic Myeloid Leukemia Patients
Brief Title: Safety and Efficacy Evaluation of Bosutinib Plus Atezolizumab in Newly Diagnosed Chronic Leukemia Adult Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study has been prematurely terminated due to the onset of 2 dose limiting toxicities in 2 patients.
Sponsor: Fundacion Espanola para la Curacion de la Leucemia Mieloide Cronica (Other)
Collaborators: Pfizer (Industry); Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEROLMC-01
Record Dates: First submitted 2021-01-19; First posted 2021-03-11 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Chronic Phase-Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — bosutinib; atezolizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bosutinib-Atezolizumab Combination (Experimental): Drugs to be administered:
  Bosutinib 400 milligram (mg)/day Oral Tablet [Bosulif 100mg oral tablets] for 1 year Atezolizumab 1680 mg/28 days [Tecentriq 840 MG in 14 ML Injection] for 1 year
  Interventions: Drug: Bosutinib 400 MG Monotherapy; Drug: Bosutinib 400 MG + Atezolizumab 840 MG in 14 ML Injection

INTERVENTIONS:
Drug: Bosutinib 400 MG Monotherapy — One cycle (28 days) only with bosutinib 400 mg/day therapy at the beginning of the trial + 12 cycles with bosutinib 400 mg/day therapy after combined therapy
  Other Names: Bosulif
Drug: Bosutinib 400 MG + Atezolizumab 840 MG in 14 ML Injection — 12 cycles with bosutinib 400 mg/day plus atezolizumab 1680 mg q4w therapy between the monotherapy bosutinib cycles
  Other Names: Bosulif + Tecentriq

SUMMARY:
The combination of bosutinib plus atezolizumab in first line treatment in newly diagnosis chronic-phase Chronic Myeloid Leukemia (CML) patients could potentially increase molecular responses and therefore treatment discontinuation probabilities in these patients. We propose an Open-Label Phase Ib/II Study of Bosutinib in Combination with Atezolizumab for the Treatment of New Diagnosis Chronic Phase-Chronic Myeloid Leukemia Patients.

DETAILED DESCRIPTION:
The combination of bosutinib and atezolizumab in first line treatment in newly diagnosis chronic-phase Chronic Myeloid Leukemia (CML) patients could potentially increase molecular responses and consequently treatment discontinuation probabilities in these patients. We would like to propose an Open-Label Phase Ib/II Study of Bosutinib in Combination with Atezolizumab for the Treatment of New Diagnosis Chronic Phase-Chronic Myeloid Leukemia Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years of age.
2. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legal representative) has been informed of all pertinent aspects of the study.
3. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
4. Newly Patient with Philadelphia chromosome positive chronic phase CML and BCR-ABL1 transcript detected at diagnosis.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
6. Adequate hepatic, renal and pancreatic function defined as:

   1. Total bilirubin within normal range or Direct bilirubin ≤ 1.5 x ULN,
   2. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) or ≤5 x ULN if attributable to liver involvement of leukemia,
7. Women of childbearing potential must have a negative pregnancy test documented prior enrollment. Women of childbearing potential and men must be using an adequate method of contraception.

Exclusion Criteria:

1. Pregnant or lactating women,
2. Participation in another clinical trial with any investigational drug within 30 days prior to study enrollment,
3. Any prior medical treatment for CML, including tyrosine kinase inhibitors (TKIs), with the exception of hydroxyurea,
4. Period of time since CML diagnosis longer than 6 months,
5. Hypersensitivity to the active substances or to any of the excipients of the bosutinib and/or atezolizumab formulations,
6. Major surgery or radiotherapy within 14 days of enrollment,
7. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease,
8. Concomitant use of or need for medications known to prolong the QTc interval,
9. Concomitant use with strong CYP3A inhibitors (ketoconazole, itraconazole, clarithromycin), moderate CYP3A inhibitors (erythromycin, fluconazole, diltiazem), or strong CYP3A inducers (rifampin, carbamazepine, phenytoin),
10. History of clinically significant or uncontrolled cardiac disease, including:

    1. Stage II to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system for heart failure.
    2. Myocardial infarction within the previous 6 months,
    3. Symptomatic cardiac arrhythmia requiring treatment,
    4. Diagnosed or suspected congenital or acquired prolonged QT history or prolonged QTc. (QTcF should not exceed 500 msec),
11. Grade III or IV fluid retention,
12. Uncontrolled hypomagnesemia or uncorrected symptomatic hypokalemia, due to potential effects on the QTc interval,
13. Uncontrolled or symptomatic hypercalcemia,
14. Recent or ongoing clinically significant gastrointestinal (GI) disorder e.g. Crohn's Disease, Ulcerative Colitis or prior total or partial gastrectomy,
15. Autoimmune or infectious active disease that require treatment,
16. CML patient not in chronic phase at diagnosis,
17. Patients with known atypical transcript. An atypical transcript is defined by the presence of any transcript in the absence of the major transcripts b3a2 (e14a2) and b2a2 (e13a2) or p210 protein,
18. Patients with known resistant mutation(s) (T315I, E255K/V, Y253H, F359C/V). It is not necessary to perform mutation tests on the patient to be included in the study if they were not previously performed,
19. Individuals with an active malignancy,
20. Known seropositivity to human immunodeficiency virus (HIV), current acute or chronic hepatitis B (hepatitis B surface-antigen positive) and/or hepatitis C.
21. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug.
22. Patients with severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Garcia, Dr., Principal Investigator — Hospital Ramon y Cajal
Locations (2):
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib-Atezolizumab Combination: Drugs to be administered:
  Bosutinib 400 MG/day Oral Tablet [Bosulif 100mg oral tablets] for 1 year Atezolizumab 1680 mg/28 days [Tecentriq 840 MG in 14 ML Injection] for 1 year
  Bosutinib 400 MG Monotherapy: One cycle (28 days) only with bosutinib 400 mg/day therapy at the beginning of the trial + 12 cycles with bosutinib 400 mg/day therapy after combined therapy
  Bosutinib 400 MG + Atezolizumab 840 MG in 14 ML Injection: 12 cycles with bosutinib 400 mg/day plus atezolizumab 1680 mg q4w therapy between the monotherapy bosutinib cycles
Period: Overall Study
Arm/Group | Bosutinib-Atezolizumab Combination
Started | 9
Completed | 4
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 9
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 47.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
BCR-ABL [Mean (Standard Deviation); unit: IS (%)] — The study's main variable is BCR-ABL ratio. The measurement of BCR-ABL1 mRNA levels were done by reverse transcription quantitative polymerase chain reaction (RT-qPCR) in peripheral blood. The results are reported as the ratio (percentage) of BCR-ABL protein (Mutated to normal ABL protein, expressed as % in the international scale [IS]) a scale developed for standardized reporting of BCR-ABL1 RNA levels. BCR-ABL1 IS = BCR-ABL1 transcript number/ABL1 transcript number × 100% × conversion coefficient (calculated for each case according to laboratory procedures and the specific calibration curve)
  IS (%) | 84.9707 (83.3527)

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Bosutinib 400 mg Daily in Combination With Atezolizumab in Participants With Chronic Myeloid Leukemia as First Line Treatments
Description: All Adverse Events, despite their severity or causal relationship with the study medication, will be reported, graded according CTCAE v5.0 and analyzed.
Time Frame: through study completion, up to 7 months
Population: The study had to be prematurely terminated due to drug toxicity; the stopping rules detailed in the protocol for safety reasons were reached. Therefore no sufficient data were obtained to conduct an efficacy analysis. No study subjects could be analysed for any of the efficacy outcomes.
Measure: Number; unit: Total No Adverse events recorded
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 9
Total No Adverse events recorded | 55

2. Secondary Outcome: To Evaluate the Molecular Response (MR) Rates
Description: Ratio of patients that reach a Molecular response
Time Frame: 7 months
Population: The study had to be prematurely terminated due to drug toxicity; the stopping rules detailed in the protocol were reached. Therefore no sufficient data were obtained to conduct the planned efficacy analysis. No study subjects could be analysed for any of the efficacy outcomes. Study has to be prematurely terminated and the analysis could not be done due to lack of data (n=0 Participants).
Groups:
- Bosutinib-Atezolizumab Combination: Drugs to be administered:
  Bosutinib 400 MG/day Oral Tablet [Bosulif 100mg oral tablets] for 1 year Atezolizumab 1680 mg/28 days [Tecentriq 840 MG in 14 ML Injection] for 1 year
  Bosutinib 400 MG Monotherapy: One cycle (28 days) only with bosutinib 400 mg/day therapy at the beginning of the trial + 12 cycles with bosutinib 400 mg/day therapy after combined therapy
  Bosutinib 400 MG + Atezolizumab 840 MG in 14 ML Injection: 12 cycles with bosutinib 400 mg/day plus atezolizumab 1680 mg q4w therapy between the monotherapy bosutinib cycles
  The study had to be prematurely terminated due to drug toxicity; the stopping rules detailed in the protocol were reached. Therefore no sufficient data were obtained to conduct the planned analysis. No study subjects could be analysed for this outcome (n=0 Participants).
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Alive
Description: Percentage of patients that remain alive at different time-points over the total number or patients
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Confirmed MR4 and MR4.5
Description: Total number of patients that reach Molecular response 4 (MR4) and Molecular Response 4.5 (MR4.5)
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

5. Secondary Outcome: The Rate of Confirmed MR4 and MR4.5
Description: Ratio of patients that reach MR4 and MR4.5
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Complete Cytogenetic Responses (CCyR)
Description: Number of patients that reach a Complete Cytogenetic Responses (CCyR)
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

7. Secondary Outcome: The Rate of Complete Cytogenetic Response (CCyR)
Description: Ratio of patients that reach a Complete Cytogenetic Responses (CCyR)
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

8. Secondary Outcome: Days to Response (CCyR, MMR, MR4, MR4.5)
Description: Number of days lasted since the beginning of the treatment upt to reach molecular response.
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

9. Secondary Outcome: The Median Time to Response (CCyR, MMR, MR4, MR4.5)
Description: Average elapsed time measured for all included patients since the beginning of the treatment up until reach measurable cytogenetic or molecular response
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

10. Secondary Outcome: Probability of Response (CCyR, MMR, MR4, MR4.5)
Description: The overall estimated probability of reaching complete cytogenetic response or molecular response MMR, MR4 or MR4.5
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Overall Surviving Patients
Description: Number of the overall surviving patients
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Progression-free Survival Patients
Description: The following events are considered disease progression:
  * Acelerated Phase.
  * Blast Crisis.
  * CML-related death.
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Failure-free Survival Patients
Description: Number of the failure-free survival patients
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Event-free Survival Patients
Description: Number of the event-free survival patients
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

15. Secondary Outcome: Phenotypical Assays of Cell Characterization
Description: Phenotypical assays of the cell characterization
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

16. Secondary Outcome: Phenotypical Assays of Differentiation, Maturation and Proliferation NK Cells Markers
Description: Phenotypical assays of the differentiation, maturation and proliferation NK cells markers
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

17. Secondary Outcome: Phenotypical Assays of CD4+ T Cells Activation Markers
Description: Phenotypical assays of the CD4+ T cells activation markers
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

18. Secondary Outcome: Phenotypical Assays of Predictive Markers of CML Relapse
Description: Phenotypical markers assessment for relapse included
  1. Cell characterization: NK cells (CD3- CD56+; CD16+ CD56+; TNFα; IFNα; Granzyme b NK-LGL cells (CD56+ CD57+), T-LGL cells (CD3+ CD57+), CD8 TCRα/β, NK markers (NKG2D, KIR2DL2/DL3/DS2, KIR2DL5B).
  2. Differentiation and maturation (NKG2A/CD16) and proliferation (NK67) markers of NK cells.
  3. CD4+ T cells activation markers: CD25 CD69 HLA-DR.
  4. Predictive markers of CML relapse: T regs (CD4+ CD25int-hi CD127low), CD8+ T cells (PD-1/PD-L1) and plasmacytoid dendritic cells (CD86+).
Time Frame: 7 months
Population: as for outcome 2
Arm/Group | Bosutinib-Atezolizumab Combination
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study Period: start (first patient enrolled) 24/02/2021 and premature end (Last patient last visit) 24/09/2021. Therefore, 7 months was the duration of this study and in this period of time when adverse event data were collected.
Description: During the study all patients reported, at least 1 AE, and at least 1 AE considered possibly, probably or definitely related to the study medication. The system most frequently affected by AE, according to SOC MedDRA organization, was, Gastrointestinal Disorders, but the most severe AEs (grade 3 and above) were those affecting the liver function. All the possibly related events were previously described as adverse reactions in the product's data sheets (Bosulif SmPC and Tencentriq SmPC).
Arm/Group | Bosutinib-Atezolizumab Combination
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib-Atezolizumab Combination (N=9)
Hepatotoxicity (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Transaminases Elevation (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosutinib-Atezolizumab Combination (N=9)
Diarrhoea (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain upper (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Hepatobiliary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Lipase increased (Metabolism and nutrition disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (2)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT04793399/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT04793399/SAP_001.pdf